CLINICAL TRIAL: NCT05865236
Title: Comparative Effect of Air Heat Versus Infra Red Heat on Pain and Wound Healling After Episiotomy
Brief Title: Comparative Effect of Air Heat Versus Infra Red Heat on Pain and Wound Healling After Vaginal Delivery Episiotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0521
Record Dates: First submitted 2023-04-18; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Episiotomy Wound
Keywords: Air Heat; Infrared Heat; Episiotomy; Kegel Exercises; Pain Relief

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical therapy Dry air heat group along with kegel exercise (Experimental): Woman should lie on the bed without panties or the sanitary Pad. Place towels under buttocks to absorb any vaginal discharge. She should lie on her back with the knees bent and feet flat. Let the vagina dry by holding a hair dryer 10 to 12 inches away from episiotomy. The dry heat will gives a soothing effect on the wound
  Interventions: Procedure: Dry air heat group + Kegal Exercises
- therapeutics execise Infra-red lamp therapy along with kegel execise (Active Comparator): The infrared the infrared lamp will be placed at distance of 45 cm away from the perineum with the heat emitted with 220 volts used for 10-15 minutes IRR is beneficial for promoting wound healing, tissue repair, and skin rejuvenation.
  Interventions: Procedure: Infra-red lamp therapy + Kegal Exercises

INTERVENTIONS:
Procedure: Infra-red lamp therapy + Kegal Exercises — The infrared the infrared lamp will be placed at distance of 45 cm away from the perineum with the heat emitted with 220 volts used for 10-15 minutes IRR is beneficial for promoting wound healing, tissue repair, and skin rejuvenation.
  Arms: therapeutics execise Infra-red lamp therapy along with kegel execise
Procedure: Dry air heat group + Kegal Exercises — Woman should lie on the bed without panties or the sanitary Pad. Place towels under buttocks to absorb any vaginal discharge. She should lie on her back with the knees bent and feet flat. Let the vagina dry by holding a hair dryer 10 to 12 inches away from episiotomy. The dry heat will gives a soothing effect on the wound
  Arms: physical therapy Dry air heat group along with kegel exercise

SUMMARY:
To become "mother" is a beautiful gift given by God to woman. Giving birth is a powerful and life changing even with a lasting impact on women and their families. Pregnancy and labor are exceptional occasions in women's lives. Post-delivery is very decisive period for compassionate woman who had under gone episiotomy which is a throbbing and disquiet procedure during this time. Episiotomy wound healing takes weeks to years depending on health conditions and treatment of the perineum itself. Episiotomy care is very essential, if neglected it can lead to severe complications like infection, wound gapping.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women
* Postnatal mothers delivered within 12-24hours.
* Have a normal vaginal delivery with episiotomy
* fand Second degree episiotomy.

Exclusion Criteria:

* Instrumental Delivery ( Forceps/ventous)
* Lower segment Cesarian section
* History of medical problem as hypertension and diabetes or anemia
* Perineal tear
* Infected wound
* Twin pregnancy

Ages: 18 Weeks to 40 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — episiotomy only check in female
Enrollment: 32 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09-02 (Estimated)

PRIMARY OUTCOMES:
REEDA Scale | 4 weeks
  REEDA Scale (Redness, Edema, Ecchymosis, Discharge and Approximation of the wound edges)

SECONDARY OUTCOMES:
NPRS Numerical Pain Rating Scale | 4 weeks
  Pain intensity is frequently measured on an 11-point pain intensity numerical rating scale (PI-NRS), where 0 = no pain and 10 = worst possible pain. The studies had similar designs and measurement instruments, including the PI-NRS, collected in a daily diary, and the standard seven- point patient global impression of change (PGIC), collected at the endpoint. The changes in the PI-NRS from baseline to the endpoint were compared to the PGIC for each subjec

CONTACTS AND LOCATIONS:
Overall Officials: mariya tariq, ms-whpt, Principal Investigator — Riphah International University
Locations (1):
- Lady Willington, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No